CLINICAL TRIAL: NCT02655731
Title: HeartLight Guided - Pure Pulmonary Vein Isolation Regardless of Concomitant Atrial Substrate
Acronym: HEURECA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cardioangiologisches Centrum Bethanien (Other)
Responsible Party: Principal Investigator, Boris Schmidt, Head of Department, Cardioangiologisches Centrum Bethanien
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FF117/2015
Record Dates: First submitted 2015-12-23; First posted 2016-01-14 (Estimated); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Other): PVI with HeartLight
  Interventions: Device: PVI with HeartLight

INTERVENTIONS:
Device: PVI with HeartLight — Catheter ablation

SUMMARY:
Aim of the present prospective, single-centre study is to determine the outcome after pure PVI using HeartLight™ in 100 patients with different extents of LA-LVA.

The latter will be assessed by an electro-anatomical voltage map using a commercial 3D mapping system (CARTO, Biosense Webster).

DETAILED DESCRIPTION:
The ablation strategy for patients with atrial fibrillation (AF) and concomitant atrial substrate (e.g. low-voltage areas; LVA) is a matter of controversy.

Results of studies investigating the impact of LVA may have been confounded by PV-to-left-atrial (LA) reconnection due to non-durable ablation. Therefore, the true contribution of LA-LVA to AF recurrences remains unknown.

Meanwhile, new ablation technologies such as the HeartLight™ laser balloon (LB) ablation system providing near complete chronic PVI rates have been developed.

Aim of the present prospective, single-centre study is to determine the outcome after pure PVI using HeartLight™ in 100 patients with different extents of LA-LVA.

The latter will be assessed by an electro-anatomical voltage map using a commercial 3D mapping system (CARTO, Biosense Webster).

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic atrial fibrillation
* Left atrial size <50mm
* Left ventricular ejection fraction <45%
* Patient is able to provide informed consent

Exclusion Criteria:

* Contraindications for PVI
* Previous PVI attempts
* Inability to be treated with oral anticoagulation
* Presence of intracardiac thrombi
* Pregnancy
* Participation in other clinical studies
* Unwilling to follow the study protocol and to attend follow-up visits

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-12; Primary Completion 2018-03-20 (Actual); Study Completion 2018-03-20 (Actual)

PRIMARY OUTCOMES:
Freedom from atrial fibrillation and atrial tachyarrhythmias | 12 months
  72h Holter-ECG recordings will be performed. In case of clinical arrhythmia symptoms event-recording will be provided.

CONTACTS AND LOCATIONS:
Overall Officials: Boris Schmidt, MD, Principal Investigator — Cardioangiologisches Centrum Bethanien
Locations (1):
- Cardioangiologisches Centrum Bethanien, Frankfurt am Main, Germany